CLINICAL TRIAL: NCT02304588
Title: Vascular Occlusive Diseases Such as Diabetic Foot Treated With Mesenchymal Stem Cell
Brief Title: Stem Cell Therapy for Patients With Vascular Occlusive Diseases Such as Diabetic Foot
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Academician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-ST-001
Record Dates: First submitted 2014-11-12; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Foot; Lower Limb Ischemia
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stem cells (Experimental): Maximal amount of MSC cells injected: 10-20*10^6 cells (up to volume of 20mL, depending on the wound size & patient weight).
  Interventions: Biological: Mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymal stem cells — 10-20 x 10^6 cells/20mL

SUMMARY:
Mesenchymal stem cells with multidirectional differentiation potential,autologous stem cell transplantation into ischemic foot, make its differentiation to form new blood capillary, improve and restore the local blood flow.

ELIGIBILITY:
Inclusion Criteria:

* the age of 30-78 years old, men and women there is no limit.
* in accordance with the ministry of health in higher medical colleges and universities teaching material the sixth edition of the annals of diabetic foot diagnostic criteria.
* with severe lower limb ischemia (defined as the resting state of ankle brachial index (ABI) 0.4-0.85, accompanied by resting or intermittent toe line.
* treatment on a voluntary basis, and sign the informed consent.

Exclusion Criteria:

* with severe heart, liver, kidney, lung function failure or general condition is very poor can't tolerate the stem cell transplant.
* clear over the past five years tumor markers in patients with malignant disease and blood levels increased significantly.
* the prodrome of acute infectious diseases.
* participated in clinical subjects within three months before test.
* adherence is poor, can not complete the course.

Ages: 30 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 months
  Frequency and severity of Adverse Events

SECONDARY OUTCOMES:
Relative Wound Area Regression of 40% or More at 6 Week | 6 week

OTHER OUTCOMES:
Reduced pain | 6 months after treatment
  Reduced pain, measured by VAS scale and use of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: xiaobing FU, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China